CLINICAL TRIAL: NCT06774430
Title: Digital Strategies to Advance Help-Seeking in Youth at Clinical High Risk for Developing Psychosis
Brief Title: Digital Strategies to Advance Help-Seeking Aim 1 and 2
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Birnbaum, Asst Professor of Clinical, Columbia University
Other Study IDs: AAAV1315 Aim 1 and 2; 1R01MH133569-01A1 (NIH)
Record Dates: First submitted 2025-01-13; First posted 2025-01-14 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Clinical High Risk; Early Psychosis; First Episode Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This proposal aims to establish a Digital Laboratory focused on advancing help-seeking and expediting treatment initiation in youth ages 12-29 who are at Clinical High-Risk (CHR) for developing psychosis. Leveraging the Health Action Process Approach (HAPA) model, this study will identify help-seeking subtypes in 25,000 youth who screen positive for psychosis-risk on Mental Health America's national online screening platform, iteratively develop and test theory and data-driven, personalized strategies to advance help-seeking using Micro-Randomized Trials and a Sequential Multiple Assignment Randomized Trial, identify the most accurate CHR screening threshold in an online environment, and link youth, when indicated, to local clinical care via Accelerating Medicines Partnership - Schizophrenia (AMP-SCZ), a NIH funded national network of CHR programs throughout the US. This academic-industry partnership aims to curate one of the largest datasets of youth with CHR, and to develop effective strategies to enhance early help-seeking, in a population where help-seeking is critical and a significant barrier to care.

DETAILED DESCRIPTION:
Aim 1: Characterize help-seeking patterns in 25,000 youth who score above Prodromal-Questionnaire (PQ-B) threshold. H1a: Youth will cluster into (1) pre-intenders (take the PQ-B and engage with educational content), (2) intenders (initiate a text exchange with a Strong365 peer navigator (3) actors (advance from texting to clinical assessment with a Strong365 clinician over phone/video) and (4) super-actors (advance from assessment to AMP-SCZ intake). Data will include online metadata (time spent online, # of resources viewed, time spent to complete the PQ-B, # of texts initiated/exchanged), self-report (demographics, symptom type and severity, PQ-B score, goals/needs, self-efficacy), and natural language. H1b (Strong365 only): Natural Language Processing (NLP) of data extracted from participant/provider interactions over text and video will identify linguistic markers of HAPA stages: intender, actor, super-actor. Models based on HAPA stages, along with behavioral features (i.e., message timing, frequency, response lag) will predict help-seeking advancement vs. disengagement. Top predictive features will be used to inform the crafting of help-seeking advancement strategies to be tested in MRTs (Aim 3).

Aim 2: To ensure that those who complete the PQ-B are directed appropriately, this study will establish the most accurate threshold for identifying CHR online. H2: Using data from population-based PQ-B screening, the investigators predict that a total distress score of 20+ will generate the highest diagnostic odds ratio with a sensitivity of at least 80% online, as determined by remote clinical assessment. For the remainder of the study, the threshold score that maximizes specificity and sensitivity will be used.

ELIGIBILITY:
Inclusion Criteria:

* Ages 12-29 years
* Living within a 50-mile radius of a US based AMP-SCZ site
* Able to complete the English language PQ-B on MHA's screening platform

Ages: 12 Years to 29 Years | Sex: All
Age Groups: Child, Adult
Study Population: Based on current MHA user demographic data, the investigators expect a high percentage of youth from low-income families (over 50% report household income below $40,000/year) who have never been in psychiatric care (65% of those who screen positive report having no mental health diagnosis). MHA visitors who complete the PQ-B are a diverse and representative sample of US youth in terms of racial, ethnic, sexual orientation, and gender identity.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Proportion of participants in each help-seeking category | 1 year
  Data from participants, including online metadata (time spent online, # of resources viewed, time spent to complete the PQ-B, # of texts initiated/exchanged), self-report (demographics, symptom type and severity, PQ-B score, goals/needs, self-efficacy), and natural language will be used to cluster participants into 4 categories: (1) Pre-intenders (take the PQ-B); (2) Intenders (initiate a text exchange with a peer navigator; (3) Actors (advance to clinical assessment); and (4) Super-actors (advance to intake).
Aim 2: Threshold score for identifying Clinical High-Risk Youth online | 1 year
  This score will be determined using data from population-based PQ-B screening. A total distress score of 20+ is predicted to generate the highest diagnostic odds ratio with a sensitivity of at least 80% online, as determined by remote clinical assessment. For the remainder of the study, a threshold score that maximizes specificity and sensitivity will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Birnbaum, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States